CLINICAL TRIAL: NCT06505616
Title: SOLFA Study: A Multicenter, Open-label, Prospective, Randomized Study to Explore the Clotting Propensity of Solacea™ Dialyser Comparing With Synthetic Membranes
Brief Title: SOLFA Study to Explore the Thrombogenicity of a Dialyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Senefro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SENEFRO SOLFA study
Record Dates: First submitted 2024-06-05; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: anticoagulation; heparin; biocompatibility; haemodialysis; haemodiafiltration; haemodialyser

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, randomized, crossover, non-masked study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asymmetric cellulose triacetate (ATA™) membrane (Solacea™, Nipro, Osaka, Japan) (Active Comparator): Patients were dialyzed with an asymmetric cellulose triacetate (ATA™) membrane (Solacea™, Nipro, Osaka, Japan). Non synthetic membrane, cellulose membrane.
  Interventions: Device: Compared the trombogenicity of the Solacea dialyzer with synthetic dialyzers after progressively decreasing heparin until discontinuing it
- Synthetic haemodialysers membranes (Active Comparator): Synthetic haemodialysis membranes habitual used in the hospitals included in the study: FXCorDiax 800™ (Fresenius MC),Polyflux 210H™ (Baxter),Revaclear 400™ (Baxter),Eliseo 19H™ (Nipro)
  Interventions: Device: Compared the trombogenicity of the Solacea dialyzer with synthetic dialyzers after progressively decreasing heparin until discontinuing it

INTERVENTIONS:
Device: Compared the trombogenicity of the Solacea dialyzer with synthetic dialyzers after progressively decreasing heparin until discontinuing it — The duration of the study was four weeks, carried out in two phases. After screening, patients were randomized to be dialyzed with the Solacea™ hemodialyzer versus the usual hemodialyzer, which in all cases had to be a synthetic membrane. In both arms, heparin was progressively decreased until it was discontinued. Afterwards the patients were crossed over to the other arm.

SUMMARY:
Prospective, multicenter, randomized, crossover, non-masked study to evaluate the impact on the thrombogenicity of the haemodialysis circuit by comparing synthetic haemodialysers against the ATA membrane of the Solacea™.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, crossover, non-masked study that included 32 patients from 4 Spanish hospitals.

The objective of the present work is to evaluate the impact on the thrombogenicity of the haemodialysis circuit by comparing synthetic haemodialysers against the ATA membrane of the Solacea™.

Study population. Patients over 18 years of age in a chronic haemodialysis program who had been on dialysis for more than three months were included. All patients provided informed consent. The study was approved by the local Ethics Committee and was conducted according to the principles of the Declaration of Helsinki. The exclusion criteria were allergies to synthetic membranes and allergies to heparin, patients receiving anticoagulant treatment, women Pregnant, breastfeeding or patients with cognitive impairment.

In each of the two phases of six consecutive two-week HD sessions, patients were dialyzed according to their usual schedule with the haemodialyser assigned after randomization (synthetic vs ATA membrane). During the six sessions of both phases, the dose of heparin was progressively reduced, 100% usual heparin dose in the first session until sixth session without heparin.

After each session, carried out a visual inspection of the venous chamber and the haemodialyser and assigned a coagulation score previously published. Dialyser score from 0 (completly clean, 0% coagulated fibers) to 4 (100% coagulated fibers). Venous chamber score from 0 (clean, without clotting) to 3 (complete oclusión, dialysis is not possible).

Demographic data and dialysis parameters were also collected. The dialyzers from 8 patients were collected at the beginning and end of each study arm and scanned with a reference non-invasive micro-CT (Computed Tomography) scanning technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients in a chronic haemodialysis program who had been on dialysis for more than three months were included.
* Patients provided informed consent.

Exclusion Criteria:

* allergies to synthetic membranes
* allergies to heparin
* patients receiving anticoagulant treatment
* women Pregnant
* breastfeeding
* patients with cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Impact on the thrombogenicity of the haemodialysis circuit by comparing dialyzers | four weeks, carried out in two phases
  The investigators measure the impact of Solacea membrane on the thrombogenicity of the haemodialysis circuit compared to other high-permeability synthetic dialysers commonly used in clinical practice.
  Heparin was progressively reduced until it was discontinued. After each session, investigators carried out a visual inspection of the venous chamber and the haemodialyser and assigned a coagulation score. In 8 patients also a scanning technique was carried out.

SECONDARY OUTCOMES:
Effect of heparin reduction or discontinuation | four weeks, carried out in two phases
  The investigators measure the effect of heparin reduction or discontinuation on vascular access haemostasis time, on dialysis efficacy by measuring KT, on percentage reduction of molecules such as myoglobin or β2-microglobulin, and in the amount of convective volume in patients in OL HDF. During the six sessions of both phases, the dose of heparin was progressively reduced until the last session without heparin. After each session, carried out a visual inspection of the venous chamber and the haemodialyser and assigned a coagulation score. In 8 patients also a scanning technique was carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Puerta, MD, Principal Investigator — University Hospital Infanta Leonor
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Claudel SE, Miles LA, Murea M. Anticoagulation in hemodialysis: A narrative review. Semin Dial. 2021 Mar;34(2):103-115. doi: 10.1111/sdi.12932. Epub 2020 Nov 1. PMID 33135208
- [Result] Davenport A. What are the anticoagulation options for intermittent hemodialysis? Nat Rev Nephrol. 2011 Jul 5;7(9):499-508. doi: 10.1038/nrneph.2011.88. PMID 21727925
- [Result] Sahota S, Rodby R. Inpatient hemodialysis without anticoagulation in adults. Clin Kidney J. 2014 Dec;7(6):552-6. doi: 10.1093/ckj/sfu114. Epub 2014 Oct 30. PMID 25859371
- [Result] Guery B, Alberti C, Servais A, Harrami E, Bererhi L, Zins B, Touam M, Joly D. Hemodialysis without systemic anticoagulation: a prospective randomized trial to evaluate 3 strategies in patients at risk of bleeding. PLoS One. 2014 May 13;9(5):e97187. doi: 10.1371/journal.pone.0097187. eCollection 2014. PMID 24825343
- [Result] Nakornchai P, Jitraree A, Homjan MC, Laykhram T, Trakarnvanich T. Comparison of citrate dialysate in pre- and post-dilution online hemodiafiltration: effect on clot formation and adequacy of dialysis in hemodialysis patients. Ren Fail. 2024 Dec;46(1):2302109. doi: 10.1080/0886022X.2024.2302109. Epub 2024 Jan 8. PMID 38189095
- [Result] Laville M, Dorval M, Fort Ros J, Fay R, Cridlig J, Nortier JL, Juillard L, Debska-Slizien A, Fernandez Lorente L, Thibaudin D, Franssen C, Schulz M, Moureau F, Loughraieb N, Rossignol P. Results of the HepZero study comparing heparin-grafted membrane and standard care show that heparin-grafted dialyzer is safe and easy to use for heparin-free dialysis. Kidney Int. 2014 Dec;86(6):1260-7. doi: 10.1038/ki.2014.225. Epub 2014 Jul 9. PMID 25007166
- [Result] Bramham K, Varrier M, Asgari E, Makanjuola D. Comparison of Tinzaparin and unfractionated heparin as anticoagulation on haemodialysis: equal safety, efficacy and economical parity. Nephron Clin Pract. 2008;110(2):c107-13. doi: 10.1159/000158561. Epub 2008 Sep 30. PMID 18824874
- [Result] Maduell F, Moreso F, Pons M, Ramos R, Mora-Macia J, Carreras J, Soler J, Torres F, Campistol JM, Martinez-Castelao A; ESHOL Study Group. High-efficiency postdilution online hemodiafiltration reduces all-cause mortality in hemodialysis patients. J Am Soc Nephrol. 2013 Feb;24(3):487-97. doi: 10.1681/ASN.2012080875. Epub 2013 Feb 14. PMID 23411788
- [Result] Blankestijn PJ, Vernooij RWM, Hockham C, Strippoli GFM, Canaud B, Hegbrant J, Barth C, Covic A, Cromm K, Cucui A, Davenport A, Rose M, Torok M, Woodward M, Bots ML; CONVINCE Scientific Committee Investigators. Effect of Hemodiafiltration or Hemodialysis on Mortality in Kidney Failure. N Engl J Med. 2023 Aug 24;389(8):700-709. doi: 10.1056/NEJMoa2304820. Epub 2023 Jun 16. PMID 37326323
- [Result] Sombolos KI, Fragia TK, Gionanlis LC, Veneti PE, Bamichas GI, Fragidis SK, Georgoulis IE, Natse TA. The anticoagulant activity of enoxaparin sodium during on-line hemodiafiltration and conventional hemodialysis. Hemodial Int. 2009 Jan;13(1):43-7. doi: 10.1111/j.1542-4758.2009.00336.x. PMID 19210277
- [Result] Vanommeslaeghe F, Josipovic I, Boone M, Dhondt A, Van Biesen W, Eloot S. A randomized cross-over study with objective quantification of the performance of an asymmetric triacetate and a polysulfone dialysis membrane using different anticoagulation strategies. Clin Kidney J. 2019 Dec 22;14(1):398-407. doi: 10.1093/ckj/sfz163. eCollection 2021 Jan. PMID 33564444
- [Derived] Puerta M, Jaldo MT, Munoz P, Martinez-Miguel P, Maduell F, Lancho C, Garcia-Herrera AL, Eloot S, de Sequera P. SOLFA study: a multicenter, open-label, prospective, randomized study to investigate the clotting propensity of asymmetric cellulose triacetate membrane compared to synthetic membranes in on line HDF. J Nephrol. 2025 Mar;38(2):697-705. doi: 10.1007/s40620-024-02197-y. Epub 2025 Jan 19. PMID 39827429